CLINICAL TRIAL: NCT00145600
Title: Risk-Adapted Therapy for Pediatric Hodgkin's Disease
Brief Title: Therapy for Pediatric Hodgkin Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HOD99; NCI-2011-03721 (Registry Identifier: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2005-09-02; First posted 2005-09-05 (Estimated); Results first posted 2013-05-07 (Estimated); Last update posted 2022-10-20 (Actual); Status verified 2022-09

CONDITIONS: Hodgkin Lymphoma
Keywords: Lymphoma; Hodgkin Disease
MeSH Terms: conditions — Hodgkin Disease; Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Unfavorable Risk, Group 2 (Experimental): Unfavorable risk, group 2 arm in patients with Hodgkin's disease (n=146)
  Interventions: Drug: 12 Week Stanford V Chemotherapy
- Favorable Risk (Experimental): Favorable Risk arm in patients with Hodgkin's Disease (n=91).
  Interventions: Drug: 4 cycles of VAMP chemotherapy
- Intermediate Risk (Experimental): Intermediate Arm in patients with Hodgkins's disease (n=46).
  Interventions: Drug: 2 alternating cycles of VAMP/COP chemotherapy
- Unfavorable Risk, Group 1 (Experimental): Unfavorable risk group 1 closed early due to excessive number of adverse events (n=13).
  Interventions: Drug: 3 alternating cycles of VAMP/COP chemotherapy

INTERVENTIONS:
Drug: 12 Week Stanford V Chemotherapy — 12 weeks of Stanford V chemotherapy plus low-dose, involved-field RT in children
  Arms: Unfavorable Risk, Group 2
Drug: 4 cycles of VAMP chemotherapy — 4 cycles of VAMP chemotherapy alone in patients who achieve a complete response after 2 cycles of VAMP chemotherapy. For patients that do not achieve a complete response after 2 cycles of VAMP, they will receive low low-dose involved field radiotherapy at the end of all chemotherapy.
  Arms: Favorable Risk
Drug: 2 alternating cycles of VAMP/COP chemotherapy — 2 alternating cycles of VAMP/COP chemotherapy (total 4 cycles of chemotherapy) plus low-dose, involved-field RT.
  Arms: Intermediate Risk
Drug: 3 alternating cycles of VAMP/COP chemotherapy — 3 alternating cycles of VAMP/COP chemotherapy (total 6 cycles of chemotherapy) plus low-dose, involved-field RT
  Arms: Unfavorable Risk, Group 1

SUMMARY:
With the success of current chemotherapy for Hodgkin's disease, the goal of this protocol is to maintain the currently successful cure rate and reduce treatment related side effects and long term toxicity. The main purpose of this study is to estimate the event free survival of patients treated with risk-adapted therapy compared to historical controls.

DETAILED DESCRIPTION:
This study will evaluate the following objectives:

Primary Objectives:

1. To evaluate the efficacy of 4 cycles of VAMP chemotherapy alone in patients with favorable risk Hodgkin's disease who achieve a complete response after 2 cycles of VAMP chemotherapy.
2. To evaluate the efficacy of 4 cycles VAMP chemotherapy plus low dose RT in patients with favorable risk Hodgkin's disease who achieve a partial response after 2 cycles of VAMP chemotherapy.
3. To evaluate the efficacy of 2 alternating cycles of VAMP/COP chemotherapy (total 4 cycles of chemotherapy) plus low-dose, involved-field RT in children with intermediate risk Hodgkin's disease.
4. To evaluate the efficacy of 12 weeks of Stanford V chemotherapy plus low-dose, involved-field RT in children with unfavorable risk Hodgkin's disease.

Secondary Objectives:

1. To evaluate patient quality of life during and after treatment from the patient and parent perspective.
2. To compare patient and parental ratings of treatment-related symptoms and patient physical, psychological, social and cognitive functioning before the first treatment (T1 - baseline); after Cycle 2 or after 8 weeks of Stanford V (T2 - Evaluate Response); after cycle 4 or after 12 weeks of Stanford V and before or on the first day of radiation (as applicable) (T3); at the conclusion of radiation or within a few days following the end of radiation (as applicable) (T4); and at 3 to 6 months after completion of therapy follow-up evaluation (T5).

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients must have histologically confirmed previously untreated Hodgkin's disease (Patients receiving limited emergent RT or steroid therapy because of cardiopulmonary decompensation or spinal cord compression will be eligible for protocol enrollment).
* Patients must be 21 years of age or younger
* Ann Arbor stages IIB-IV
* No prior treatment.
* No pregnant or lactating women.
* Signed informed consent
* If re-evaluation of a patient's disease shows favorable risk features or intermediate risk features, the patient will be removed from the HOD99 study and consented to the respective HOD08 or HOD05 study.

Inclusion: treatment of favorable risk features:

* Ann Arbor IA or IIA with:

  1. Non-bulky mediastinal disease (<33% mediastinal to thoracic ratio on chest x ray)
  2. Ann Arbor stage IA or IIA with any of the following features: (1) "E" lesions (s), (2) 3 or more nodal sites involved, (3) Bulky mediastinal adenopathy (mediastinal mass to thoracic cavity ratio 33% or greater by chest radiograph)

     Inclusion: unfavorable risk features:
* Stage must be classified as one of the following:

  1. Ann Arbor stage IIB, IIIB, or any IV

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 296 (Actual)
Dates: Start 2000-03-02 (Actual); Primary Completion 2012-05-31 (Actual); Study Completion 2021-11-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jamie Flerlage, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (5):
- United States (5):
  - Stanford University, Palo Alto, California
  - Maine Children's Cancer Program, Portland, Maine
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - St. Jude Children's Research Hospital, Memphis, Tennessee

REFERENCES:
- [Derived] Metzger ML, Weinstein HJ, Hudson MM, Billett AL, Larsen EC, Friedmann A, Howard SC, Donaldson SS, Krasin MJ, Kun LE, Marcus KJ, Yock TI, Tarbell N, Billups CA, Wu J, Link MP. Association between radiotherapy vs no radiotherapy based on early response to VAMP chemotherapy and survival among children with favorable-risk Hodgkin lymphoma. JAMA. 2012 Jun 27;307(24):2609-16. doi: 10.1001/jama.2012.5847. PMID 22735430
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 296 patients were enrolled from 5 institutions between March 2000 and May 2011.
Groups:
- Favorable Risk: Ann Arbor stage IA or IIA with:
  1. Non-bulky mediastinal disease (<33% mediastinal to thoracic ratio on chest x-ray)
  2. < 3 nodal regions involved on the same side of the diaphragm
  3. No extranodal extension of disease
- Intermediate Risk: Stage must be classified as one of the following:
  1. Ann Arbor stage IB and IIIA
  2. Ann Arbor stage IA or IIA with ANY of the following features: (1) extranodal extension of disease lesion(s), (2) 3 or more nodal sites involved, (3) Bulky mediastinal adenopathy (mediastinal mass to thoracic cavity ratio 33% or greater by chest radiograph)
- Unfavorable Risk, Group 2: Stage must be classified as one of the following:
  a. Ann Arbor stage IIB, IIIB, or any IV
Period: Overall Study
Arm/Group | Favorable Risk | Intermediate Risk | Unfavorable Risk, Group 1 | Unfavorable Risk, Group 2
Started | 91 | 46 | 13 | 146
Completed | 83 | 36 | 8 | 130
Not Completed | 8 | 10 | 5 | 16
Not completed — Death | 1 | 2 | 2 | 6
Not completed — Ineligible | 3 | 0 | 1 | 5
Not completed — Lost to Follow-up | 2 | 6 | 2 | 4
Not completed — Noncompliance | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 2 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Favorable Risk | Intermediate Risk | Unfavorable Risk, Group 1 | Unfavorable Risk, Group 2 | Total
Number analyzed (Participants) | 91 | 46 | 13 | 146 | 296
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 84 | 36 | 11 | 122 | 253
  Between 18 and 65 years | 7 | 10 | 2 | 24 | 43
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.08 (3.91) | 15.35 (3.28) | 14.85 (3.21) | 15.06 (3.37) | 14.48 (3.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 26 | 5 | 80 | 143
  Male | 59 | 20 | 8 | 66 | 153

OUTCOME MEASURES:

1. Primary Outcome: Event-free Survival Probability by Risk Group
Description: Event-free survival (EFS) is based on the time from protocol enrollment to the occurrence of first event (relapse or progressive disease, subsequent malignancy, or death from any cause). Patients not experiencing an event are censored at their last follow-up date. Event-free Survival Probability will be estimated by Kaplan-Meier (KM) method with a 95% confidence interval calculated using the Greenwood's formula.
Time Frame: Median 6.4 year follow-up
Population: Nine patients were ineligible for analysis.
Measure: Number (95% Confidence Interval); unit: probability of 5 yr. event free survival
Arm/Group | Favorable Risk | Intermediate Risk | Unfavorable Risk, Group 1 | Unfavorable Risk, Group 2
Number analyzed (Participants) | 88 | 46 | 12 | 141
probability of 5 yr. event free survival | 0.886 [0.820 to 0.953] | 0.844 [0.739 to 0.950] | 0.667 [0.400 to 0.933] | 0.793 [0.726 to 0.860]
Statistical Analysis 1: Comparison: Favorable Risk; Test type: Superiority or Other; KM Event-free survival estimate = 0.886, 95% CI 2-sided [0.820 to 0.953]
Statistical Analysis 2: Comparison: Intermediate Risk; Test type: Superiority or Other; KM event-free survival estimate = 0.844, 95% CI 2-sided [0.739 to 0.950]
Statistical Analysis 3: Comparison: Unfavorable Risk, Group 1; Test type: Superiority or Other; KM event-free survival estimate = 0.667, 95% CI 2-sided [0.400 to 0.933]
Statistical Analysis 4: Comparison: Unfavorable Risk, Group 2; Test type: Superiority or Other; KM event-free survival estimate = 0.793, 95% CI 2-sided [0.726 to 0.860]

2. Secondary Outcome: Correlation of Agreement Between Patient Physical QoL and Parent Proxy Physical QoL at Multiple Time Points.
Description: Assess and compare the patient reported and parent proxy physical quality of life across multiple time points using the Peds Quality of Life version 4. Assessment was performed across all risk groups. The QL scoring is a 5-point Likert scale from 0 (never) to 4 (almost always). Scores are transformed on a scale from 0 to 100. Items are reverse scored and linearly transformed to a 0-100 scale as follows: 0=100, 1=75, 2=50, 3=25, and 4=0. Total score is the sum of all items over the number of items answered on all scales. The higher the score, the better the quality of life.
Time Frame: At Diagnosis (T1), completion of 2 cycles of chemotherapy (T2), completion of 4 cycles of chemotherapy (T3), and 3-6 months after the completion of therapy (T5).
Population: Each participating institution made the decision to complete or not complete the QoL secondary aim. Of 296 eligible participants, 178 participated in the QoL assessment. For each time point, a matching participant and parent were required to evaluate each QoL question. We had some missing data and those over 18 years did not have parent proxy.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Patient At Diagnosis (T1); Parent At Diagnosis (T1): Patients and parents were assessed for quality of life at Diagnosis (T1).
- Patient Completion of 2 Cycles of Chemotherapy (T2); Parent Completion of 2 Cycles of Chemotherapy (T2): Patients and parents were assessed for quality of life at completion of 2 cycles of chemotherapy (T2).
- Patient Completion of 4 Cycles of Chemotherapy (T3); Parent Completion of 4 Cycles of Chemotherapy (T3): Patients and parents were assessed for quality of life at completion of 4 cycles of chemotherapy (T3).
- Patient 3-6 Months After the Completion of Therapy (T5); Parent 3-6 Months After the Completion of Therapy (T5): Patients and parents were assessed for quality of life at 3-6 months after the completion of therapy (T5).
Arm/Group | Patient At Diagnosis (T1) | Parent At Diagnosis (T1) | Patient Completion of 2 Cycles of Chemotherapy (T2) | Parent Completion of 2 Cycles of Chemotherapy (T2) | Patient Completion of 4 Cycles of Chemotherapy (T3) | Parent Completion of 4 Cycles of Chemotherapy (T3) | Patient 3-6 Months After the Completion of Therapy (T5) | Parent 3-6 Months After the Completion of Therapy (T5)
Number analyzed (Participants) | 152 | 152 | 145 | 145 | 139 | 139 | 109 | 109
units on a scale | 77.2 (21.4) | 73.9 (24.5) | 72.3 (20.2) | 65.4 (21.9) | 74.7 (20.9) | 66.5 (21) | 84.5 (16.6) | 78.6 (22.7)
Statistical Analysis 1: Comparison: Patient At Diagnosis (T1) vs Parent At Diagnosis (T1); Test type: Superiority or Other; p = 0.3097, Wilcoxon signed rank test
Statistical Analysis 2: Comparison: Patient At Diagnosis (T1) vs Parent At Diagnosis (T1); Test type: Superiority or Other; p < 0.0001, Spearman Correlation Coefficients; Spearman Correlation Coefficients = 0.60
Statistical Analysis 3: Comparison: Patient Completion of 2 Cycles of Chemotherapy (T2) vs Parent Completion of 2 Cycles of Chemotherapy (T2); Test type: Superiority or Other; p < 0.0001, Wilcoxon signed rank test
Statistical Analysis 4: Comparison: Patient Completion of 2 Cycles of Chemotherapy (T2) vs Parent Completion of 2 Cycles of Chemotherapy (T2); Test type: Superiority or Other; p < 0.0001, Spearman Correlation Coefficients; Spearman Correlation Coefficients = 0.50
Statistical Analysis 5: Comparison: Patient Completion of 4 Cycles of Chemotherapy (T3) vs Parent Completion of 4 Cycles of Chemotherapy (T3); Test type: Superiority or Other; p < 0.0001, Wilcoxon signed rank test
Statistical Analysis 6: Comparison: Patient Completion of 4 Cycles of Chemotherapy (T3) vs Parent Completion of 4 Cycles of Chemotherapy (T3); Test type: Superiority or Other; p < 0.0001, Spearman Correlation Coefficients; Spearman Correlation Coefficients = 0.37
Statistical Analysis 7: Comparison: Patient 3-6 Months After the Completion of Therapy (T5) vs Parent 3-6 Months After the Completion of Therapy (T5); Test type: Superiority or Other; p = 0.0197, Wilcoxon signed rank test
Statistical Analysis 8: Comparison: Patient 3-6 Months After the Completion of Therapy (T5) vs Parent 3-6 Months After the Completion of Therapy (T5); Test type: Superiority or Other; p < 0.0001, Spearman Correlation Coefficients; Spearman Correlation Coefficients = 0.51

3. Secondary Outcome: Correlation of Agreement Between Patient Emotional QoL and Parent Proxy Emotional QoL at Multiple Time Points.
Description: Assess and compare the patient reported and parent proxy emotional quality of life across multiple time points using the Peds Quality of Life version 4. Assessment was performed across all risk groups. The QL scoring is a 5-point Likert scale from 0 (never) to 4 (almost always). Scores are transformed on a scale from 0 to 100. Items are reverse scored and linearly transformed to a 0-100 scale as follows: 0=100, 1=75, 2=50, 3=25, and 4=0. Total score is the sum of all items over the number of items answered on all scales. The higher the score, the better the quality of life.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patient At Diagnosis (T1) | Parent At Diagnosis (T1) | Patient Completion of 2 Cycles of Chemotherapy (T2) | Parent Completion of 2 Cycles of Chemotherapy (T2) | Patient Completion of 4 Cycles of Chemotherapy (T3) | Parent Completion of 4 Cycles of Chemotherapy (T3) | Patient 3-6 Months After the Completion of Therapy (T5) | Parent 3-6 Months After the Completion of Therapy (T5)
Number analyzed (Participants) | 151 | 151 | 146 | 146 | 139 | 139 | 110 | 110
units on a scale | 68.4 (18.1) | 62.3 (20.1) | 70.7 (20.5) | 64 (18.3) | 74.1 (20.4) | 65.7 (20.2) | 78.5 (21.3) | 77.1 (19.5)
Statistical Analysis 1: Comparison: Patient At Diagnosis (T1) vs Parent At Diagnosis (T1); Test type: Superiority or Other; p < 0.0001, Wilcoxon signed rank test
Statistical Analysis 2: Comparison: Patient At Diagnosis (T1) vs Parent At Diagnosis (T1); Test type: Superiority or Other; p < 0.0001, Spearman Correlation Coefficients; Spearman Correlation Coefficients = 0.46
Statistical Analysis 3: Comparison: Patient Completion of 2 Cycles of Chemotherapy (T2) vs Parent Completion of 2 Cycles of Chemotherapy (T2); Test type: Superiority or Other; p = 0.0001, Wilcoxon signed rank test
Statistical Analysis 4: Comparison: Patient Completion of 2 Cycles of Chemotherapy (T2) vs Parent Completion of 2 Cycles of Chemotherapy (T2); Test type: Superiority or Other; p < 0.0001, Spearman Correlation Coefficients; Spearman Correlation Coefficients = 0.41
Statistical Analysis 5: Comparison: Patient Completion of 4 Cycles of Chemotherapy (T3) vs Parent Completion of 4 Cycles of Chemotherapy (T3); Test type: Superiority or Other; p < 0.0001, Wilcoxon signed rank test
Statistical Analysis 6: Comparison: Patient Completion of 4 Cycles of Chemotherapy (T3) vs Parent Completion of 4 Cycles of Chemotherapy (T3); Test type: Superiority or Other; p < 0.0001, Spearman Correlation Coefficients; Spearman Correlation Coefficients = 0.42
Statistical Analysis 7: Comparison: Patient 3-6 Months After the Completion of Therapy (T5) vs Parent 3-6 Months After the Completion of Therapy (T5); Test type: Superiority or Other; p = 0.3624, Wilcoxon signed rank test
Statistical Analysis 8: Comparison: Patient 3-6 Months After the Completion of Therapy (T5) vs Parent 3-6 Months After the Completion of Therapy (T5); Test type: Superiority or Other; p < 0.0001, Spearman Correlation Coefficients; Spearman Correlation Coefficients = 0.52

4. Secondary Outcome: Correlation of Agreement Between Patient Social QoL and Parent Proxy Social QoL at Multiple Time Points.
Description: Assess and compare the patient reported and parent proxy social quality of life across multiple time points using the Peds Quality of Life version 4. Assessment was performed across all risk groups. The QL scoring is a 5-point Likert scale from 0 (never) to 4 (almost always). Scores are transformed on a scale from 0 to 100. Items are reverse scored and linearly transformed to a 0-100 scale as follows: 0=100, 1=75, 2=50, 3=25, and 4=0. Total score is the sum of all items over the number of items answered on all scales. The higher the score, the better the quality of life.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patient At Diagnosis (T1) | Parent At Diagnosis (T1) | Patient Completion of 2 Cycles of Chemotherapy (T2) | Parent Completion of 2 Cycles of Chemotherapy (T2) | Patient Completion of 4 Cycles of Chemotherapy (T3) | Parent Completion of 4 Cycles of Chemotherapy (T3) | Patient 3-6 Months After the Completion of Therapy (T5) | Parent 3-6 Months After the Completion of Therapy (T5)
Number analyzed (Participants) | 151 | 151 | 144 | 144 | 138 | 138 | 110 | 110
units on a scale | 87.2 (16) | 83 (20.2) | 87.2 (14.5) | 81.4 (17.8) | 88.2 (12.9) | 82.2 (16.2) | 91.5 (13.2) | 85.8 (17.4)
Statistical Analysis 1: Comparison: Patient At Diagnosis (T1) vs Parent At Diagnosis (T1); Test type: Superiority or Other; p = 0.0254, Wilcoxon signed rank test
Statistical Analysis 2: Comparison: Patient At Diagnosis (T1) vs Parent At Diagnosis (T1); Test type: Superiority or Other; p < 0.0001, Spearman Correlation Coefficients; Spearman Correlation Coefficients = 0.44
Statistical Analysis 3: Comparison: Patient Completion of 2 Cycles of Chemotherapy (T2) vs Parent Completion of 2 Cycles of Chemotherapy (T2); Test type: Superiority or Other; p = 0.0004, Wilcoxon signed rank test
Statistical Analysis 4: Comparison: Patient Completion of 2 Cycles of Chemotherapy (T2) vs Parent Completion of 2 Cycles of Chemotherapy (T2); Test type: Superiority or Other; p = 0.0001, Spearman Correlation Coefficients; Spearman Correlation Coefficients = 0.32
Statistical Analysis 5: Comparison: Patient Completion of 4 Cycles of Chemotherapy (T3) vs Parent Completion of 4 Cycles of Chemotherapy (T3); Test type: Superiority or Other; p < 0.0001, Wilcoxon Correlation Coefficients
Statistical Analysis 6: Comparison: Patient Completion of 4 Cycles of Chemotherapy (T3) vs Parent Completion of 4 Cycles of Chemotherapy (T3); Test type: Superiority or Other; p < 0.0001, Spearman Correlation Coefficients; Spearman Correlation Coefficients = 0.39
Statistical Analysis 7: Comparison: Patient 3-6 Months After the Completion of Therapy (T5) vs Parent 3-6 Months After the Completion of Therapy (T5); Test type: Superiority or Other; p = 0.0014, Wilcoxon signed rank test
Statistical Analysis 8: Comparison: Patient 3-6 Months After the Completion of Therapy (T5) vs Parent 3-6 Months After the Completion of Therapy (T5); Test type: Superiority or Other; p = 0.0061, Spearman Correlation Coefficients; Spearman Correlation Coefficients = 0.26

5. Secondary Outcome: Correlation of Agreement Between Patient School QoL and Parent Proxy School QoL at Multiple Time Points.
Description: Assess and compare the patient reported and parent proxy school quality of life across multiple time points using the Peds Quality of Life version 4. Assessment was performed across all risk groups. The QL scoring is a 5-point Likert scale from 0 (never) to 4 (almost always). Scores are transformed on a scale from 0 to 100. Items are reverse scored and linearly transformed to a 0-100 scale as follows: 0=100, 1=75, 2=50, 3=25, and 4=0. Total score is the sum of all items over the number of items answered on all scales. The higher the score, the better the quality of life.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patient At Diagnosis (T1) | Parent At Diagnosis (T1) | Patient Completion of 2 Cycles of Chemotherapy (T2) | Parent Completion of 2 Cycles of Chemotherapy (T2) | Patient Completion of 4 Cycles of Chemotherapy (T3) | Parent Completion of 4 Cycles of Chemotherapy (T3) | Patient 3-6 Months After the Completion of Therapy (T5) | Parent 3-6 Months After the Completion of Therapy (T5)
Number analyzed (Participants) | 129 | 129 | 114 | 114 | 106 | 106 | 95 | 95
units on a scale | 69.6 (18) | 66.2 (22.1) | 67.2 (20.6) | 66.7 (21.8) | 69 (21.6) | 66.7 (21.6) | 78.6 (18.3) | 76.5 (20)
Statistical Analysis 1: Comparison: Patient At Diagnosis (T1) vs Parent At Diagnosis (T1); Test type: Superiority or Other; p = 0.0687, Wilcoxon signed rank test
Statistical Analysis 2: Comparison: Patient At Diagnosis (T1) vs Parent At Diagnosis (T1); Test type: Superiority or Other; p < 0.0001, Spearman Correlation Coefficient; Spearman Correlation Coefficients = 0.65
Statistical Analysis 3: Comparison: Patient Completion of 2 Cycles of Chemotherapy (T2) vs Parent Completion of 2 Cycles of Chemotherapy (T2); Test type: Superiority or Other; p = 0.9478, Wilcoxon signed rank test
Statistical Analysis 4: Comparison: Patient Completion of 2 Cycles of Chemotherapy (T2) vs Parent Completion of 2 Cycles of Chemotherapy (T2); Test type: Superiority or Other; p < 0.0001, Spearman Correlation Coefficients; Spearman Correlation Coefficients = 0.42
Statistical Analysis 5: Comparison: Patient Completion of 4 Cycles of Chemotherapy (T3) vs Parent Completion of 4 Cycles of Chemotherapy (T3); Test type: Superiority or Other; p = 0.2999, Wilcoxon signed rank test
Statistical Analysis 6: Comparison: Patient Completion of 4 Cycles of Chemotherapy (T3) vs Parent Completion of 4 Cycles of Chemotherapy (T3); Test type: Superiority or Other; p < 0.0001, Spearman Correlation Coefficients; Spearman Correlation Coefficients = 0.49
Statistical Analysis 7: Comparison: Patient 3-6 Months After the Completion of Therapy (T5) vs Parent 3-6 Months After the Completion of Therapy (T5); Test type: Superiority or Other; p = 0.3121, Wilcoxon signed rank test
Statistical Analysis 8: Comparison: Patient 3-6 Months After the Completion of Therapy (T5) vs Parent 3-6 Months After the Completion of Therapy (T5); Test type: Superiority or Other; p < 0.0001, Spearman Correlation Coefficients; Spearman Correlation Coefficients = 0.52

6. Secondary Outcome: Correlation of Agreement Between Patient Psychosocial QoL and Parent Proxy Psychosocial QoL at Multiple Time Points.
Description: Assess and compare the patient reported and parent proxy psychosocial quality of life across multiple time points using the Peds Quality of Life version 4. Assessment was performed across all risk groups. The QL scoring is a 5-point Likert scale from 0 (never) to 4 (almost always). Scores are transformed on a scale from 0 to 100. Items are reverse scored and linearly transformed to a 0-100 scale as follows: 0=100, 1=75, 2=50, 3=25, and 4=0. Total score is the sum of all items over the number of items answered on all scales. The higher the score, the better the quality of life.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patient At Diagnosis (T1) | Parent At Diagnosis (T1) | Patient Completion of 2 Cycles of Chemotherapy (T2) | Parent Completion of 2 Cycles of Chemotherapy (T2) | Patient Completion of 4 Cycles of Chemotherapy (T3) | Parent Completion of 4 Cycles of Chemotherapy (T3) | Patient 3-6 Months After the Completion of Therapy (T5) | Parent 3-6 Months After the Completion of Therapy (T5)
Number analyzed (Participants) | 129 | 129 | 114 | 114 | 106 | 106 | 95 | 95
units on a scale | 75.7 (13.5) | 71.3 (16.4) | 75.1 (15) | 71.1 (15.3) | 77.5 (15.1) | 72.3 (15.9) | 83.1 (14.7) | 80.7 (15.9)
Statistical Analysis 1: Comparison: Patient At Diagnosis (T1) vs Parent At Diagnosis (T1); Test type: Superiority or Other; p = 0.0014, Wilcoxon signed rank test
Statistical Analysis 2: Comparison: Patient At Diagnosis (T1) vs Parent At Diagnosis (T1); Test type: Superiority or Other; p < 0.0001, Spearman Correlation Coefficients; Spearman Correlation Coefficients = 0.57
Statistical Analysis 3: Comparison: Patient Completion of 2 Cycles of Chemotherapy (T2) vs Parent Completion of 2 Cycles of Chemotherapy (T2); Test type: Superiority or Other; p = 0.0282, Wilcoxon signed rank test
Statistical Analysis 4: Comparison: Patient Completion of 2 Cycles of Chemotherapy (T2) vs Parent Completion of 2 Cycles of Chemotherapy (T2); Test type: Superiority or Other; p = 0.0002, Spearman Correlation Coefficients; Spearman Correlation Coefficients = 0.35
Statistical Analysis 5: Comparison: Patient Completion of 4 Cycles of Chemotherapy (T3) vs Parent Completion of 4 Cycles of Chemotherapy (T3); Test type: Superiority or Other; p = 0.0038, Wilcoxon signed rank test
Statistical Analysis 6: Comparison: Patient Completion of 4 Cycles of Chemotherapy (T3) vs Parent Completion of 4 Cycles of Chemotherapy (T3); Test type: Superiority or Other; p < 0.0001, Spearman Correlation Coefficients; Spearman Correlation Coefficients = 0.43
Statistical Analysis 7: Comparison: Patient 3-6 Months After the Completion of Therapy (T5) vs Parent 3-6 Months After the Completion of Therapy (T5); Test type: Superiority or Other; p = 0.1474, Wilcoxon signed rank test
Statistical Analysis 8: Comparison: Patient 3-6 Months After the Completion of Therapy (T5) vs Parent 3-6 Months After the Completion of Therapy (T5); Test type: Superiority or Other; p < 0.0001, Spearman Correlation Coefficients; Spearman Correlation Coefficients = 0.49

7. Secondary Outcome: Correlation of Agreement Between Patient Peds QL4 (Composite) QoL and Parent Proxy Peds QL4 (Composite) QoL at Multiple Time Points.
Description: Assess and compare the patient reported and parent proxy Peds QL4 (composite) quality of life across multiple time points using the Peds Quality of Life version 4. Assessment was performed across all risk groups. The QL scoring is a 5-point Likert scale from 0 (never) to 4 (almost always). Scores are transformed on a scale from 0 to 100. Items are reverse scored and linearly transformed to a 0-100 scale as follows: 0=100, 1=75, 2=50, 3=25, and 4=0. Total score is the sum of all items over the number of items answered on all scales. The higher the score, the better the quality of life.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patient At Diagnosis (T1) | Parent At Diagnosis (T1) | Patient Completion of 2 Cycles of Chemotherapy (T2) | Parent Completion of 2 Cycles of Chemotherapy (T2) | Patient Completion of 4 Cycles of Chemotherapy (T3) | Parent Completion of 4 Cycles of Chemotherapy (T3) | Patient 3-6 Months After the Completion of Therapy (T5) | Parent 3-6 Months After the Completion of Therapy (T5)
Number analyzed (Participants) | 129 | 129 | 113 | 113 | 106 | 106 | 94 | 94
units on a scale | 76.2 (14.9) | 72.4 (17.7) | 74.2 (15.4) | 69.3 (16.2) | 77 (15.1) | 70.6 (16.1) | 84 (13.7) | 80.7 (16.2)
Statistical Analysis 1: Comparison: Patient At Diagnosis (T1) vs Parent At Diagnosis (T1); Test type: Superiority or Other; p = 0.0281, Wilcoxon signed rank test
Statistical Analysis 2: Comparison: Patient At Diagnosis (T1) vs Parent At Diagnosis (T1); Test type: Superiority or Other; p < 0.0001, Spearman Correlation Coefficients; Spearman Correlation Coefficients = 0.63
Statistical Analysis 3: Comparison: Patient Completion of 2 Cycles of Chemotherapy (T2) vs Parent Completion of 2 Cycles of Chemotherapy (T2); Test type: Superiority or Other; p = 0.0050, Wilcoxon signed rank test
Statistical Analysis 4: Comparison: Patient Completion of 2 Cycles of Chemotherapy (T2) vs Parent Completion of 2 Cycles of Chemotherapy (T2); Test type: Superiority or Other; p < 0.0001, Spearman Correlation Coefficients; Spearman Correlation Coefficients = 0.45
Statistical Analysis 5: Comparison: Patient Completion of 4 Cycles of Chemotherapy (T3) vs Parent Completion of 4 Cycles of Chemotherapy (T3); Test type: Superiority or Other; p = 0.0005, Wilcoxon signed rank test
Statistical Analysis 6: Comparison: Patient Completion of 4 Cycles of Chemotherapy (T3) vs Parent Completion of 4 Cycles of Chemotherapy (T3); Test type: Superiority or Other; p = 0.0001, Spearman Correlation Coefficients; Spearman Correlation Coefficients = 0.37
Statistical Analysis 7: Comparison: Patient 3-6 Months After the Completion of Therapy (T5) vs Parent 3-6 Months After the Completion of Therapy (T5); Test type: Superiority or Other; p = 0.0552, Wilcoxon signed rank test
Statistical Analysis 8: Comparison: Patient 3-6 Months After the Completion of Therapy (T5) vs Parent 3-6 Months After the Completion of Therapy (T5); Test type: Superiority or Other; p < 0.0001, Spearman Correlation Coefficients; Spearman Correlation Coefficients = 0.54

8. Secondary Outcome: Correlation of Agreement Between Patient Pain and Hurt QoL and Parent Proxy Pain and Hurt QoL at Multiple Time Points.
Description: Assess and compare the patient reported and parent proxy pain and hurt quality of life across multiple time points using the Peds Quality of Life version 3. Assessment was performed across all risk groups. The QL scoring is a 5-point Likert scale from 0 (never) to 4 (almost always). Scores are transformed on a scale from 0 to 100. Items are reverse scored and linearly transformed to a 0-100 scale as follows: 0=100, 1=75, 2=50, 3=25, and 4=0. Total score is the sum of all items over the number of items answered on all scales. The higher the score, the better the quality of life.
Time Frame: At completion of 2 cycles of chemotherapy (T2), completion of 4 cycles of chemotherapy (T3), and 3-6 months after the completion of therapy (T5).
Population: Of 296 eligible, 178 participated in QoL assessment. For each time point, a matching participant and parent were required to evaluate each QoL question. We had some missing data and those over 18 years did not have parent proxy. Peds QL3 is not completed at T1 for newly diagnosed patients, because it measures symptoms over the prior month.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patient Completion of 2 Cycles of Chemotherapy (T2) | Parent Completion of 2 Cycles of Chemotherapy (T2) | Patient Completion of 4 Cycles of Chemotherapy (T3) | Parent Completion of 4 Cycles of Chemotherapy (T3) | Patient 3-6 Months After the Completion of Therapy (T5) | Parent 3-6 Months After the Completion of Therapy (T5)
Number analyzed (Participants) | 143 | 143 | 131 | 131 | 106 | 106
units on a scale | 67.7 (25.2) | 57.3 (24.6) | 69.4 (26.4) | 60.2 (25.7) | 83.4 (23.4) | 77 (23.7)
Statistical Analysis 1: Comparison: Patient Completion of 2 Cycles of Chemotherapy (T2) vs Parent Completion of 2 Cycles of Chemotherapy (T2); Test type: Superiority or Other; p < 0.0001, Wilcoxon signed rank test
Statistical Analysis 2: Comparison: Patient Completion of 2 Cycles of Chemotherapy (T2) vs Parent Completion of 2 Cycles of Chemotherapy (T2); Test type: Superiority or Other; p < 0.0001, Spearman Correlation Coefficients; Spearman Correlation Coefficients = 0.53
Statistical Analysis 3: Comparison: Patient Completion of 4 Cycles of Chemotherapy (T3) vs Parent Completion of 4 Cycles of Chemotherapy (T3); Test type: Superiority or Other; p < 0.0001, Wilcoxan signed rank test
Statistical Analysis 4: Comparison: Patient Completion of 4 Cycles of Chemotherapy (T3) vs Parent Completion of 4 Cycles of Chemotherapy (T3); Test type: Superiority or Other; p < 0.0001, Spearman Correlation Coefficients; Spearman Correlation Coefficients = 0.68
Statistical Analysis 5: Comparison: Patient 3-6 Months After the Completion of Therapy (T5) vs Parent 3-6 Months After the Completion of Therapy (T5); Test type: Superiority or Other; p = 0.0017, Wilcoxon signed rank test
Statistical Analysis 6: Comparison: Patient 3-6 Months After the Completion of Therapy (T5) vs Parent 3-6 Months After the Completion of Therapy (T5); Test type: Superiority or Other; p < 0.0001, Spearman Correlation Coefficients; Spearman Correlation Coefficients = 0.50

9. Secondary Outcome: Correlation of Agreement Between Patient Nausea QoL and Parent Proxy Nausea QoL at Multiple Time Points.
Description: Assess and compare the patient reported and parent proxy nausea quality of life across multiple time points using the Peds Quality of Life version 3. Assessment was performed across all risk groups. The QL scoring is a 5-point Likert scale from 0 (never) to 4 (almost always). Scores are transformed on a scale from 0 to 100. Items are reverse scored and linearly transformed to a 0-100 scale as follows: 0=100, 1=75, 2=50, 3=25, and 4=0. Total score is the sum of all items over the number of items answered on all scales. The higher the score, the better the quality of life.
Time Frame: as for outcome 8
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patient Completion of 2 Cycles of Chemotherapy (T2) | Parent Completion of 2 Cycles of Chemotherapy (T2) | Patient Completion of 4 Cycles of Chemotherapy (T3) | Parent Completion of 4 Cycles of Chemotherapy (T3) | Patient 3-6 Months After the Completion of Therapy (T5) | Parent 3-6 Months After the Completion of Therapy (T5)
Number analyzed (Participants) | 142 | 142 | 131 | 131 | 101 | 101
units on a scale | 60.7 (22.5) | 58.6 (22) | 59.7 (24.9) | 57.7 (23.8) | 75 (22.6) | 78.9 (22.9)
Statistical Analysis 1: Comparison: Patient Completion of 2 Cycles of Chemotherapy (T2) vs Parent Completion of 2 Cycles of Chemotherapy (T2); Test type: Superiority or Other; p = 0.2758, Wilcoxon signed rank test
Statistical Analysis 2: Comparison: Patient Completion of 2 Cycles of Chemotherapy (T2) vs Parent Completion of 2 Cycles of Chemotherapy (T2); Test type: Superiority or Other; p < 0.0001, Spearman Correlation Coefficients; Spearman Correlation Coefficients = 0.60
Statistical Analysis 3: Comparison: Patient Completion of 4 Cycles of Chemotherapy (T3) vs Parent Completion of 4 Cycles of Chemotherapy (T3); Test type: Superiority or Other; p = 0.1731, Wilcoxon signed rank test
Statistical Analysis 4: Comparison: Patient Completion of 4 Cycles of Chemotherapy (T3) vs Parent Completion of 4 Cycles of Chemotherapy (T3); Test type: Superiority or Other; p < 0.0001, Spearman Correlation Coefficients; Spearman Correlation Coefficients = 0.60
Statistical Analysis 5: Comparison: Patient 3-6 Months After the Completion of Therapy (T5) vs Parent 3-6 Months After the Completion of Therapy (T5); Test type: Superiority or Other; p = 0.0846, Wilcoxon signed rank test
Statistical Analysis 6: Comparison: Patient 3-6 Months After the Completion of Therapy (T5) vs Parent 3-6 Months After the Completion of Therapy (T5); Test type: Superiority or Other; p < 0.0001, Spearman Correlation Coefficients; Spearman Correlation Coefficients = 0.46

10. Secondary Outcome: Correlation of Agreement Between Patient Procedural Anxiety QoL and Parent Proxy Procedural Anxiety QoL at Multiple Time Points.
Description: Assess and compare the patient reported and parent proxy procedural anxiety quality of life across multiple time points using the Peds Quality of Life version 3. Assessment was performed across all risk groups. The QL scoring is a 5-point Likert scale from 0 (never) to 4 (almost always). Scores are transformed on a scale from 0 to 100. Items are reverse scored and linearly transformed to a 0-100 scale as follows: 0=100, 1=75, 2=50, 3=25, and 4=0. Total score is the sum of all items over the number of items answered on all scales. The higher the score, the better the quality of life.
Time Frame: as for outcome 8
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patient Completion of 2 Cycles of Chemotherapy (T2) | Parent Completion of 2 Cycles of Chemotherapy (T2) | Patient Completion of 4 Cycles of Chemotherapy (T3) | Parent Completion of 4 Cycles of Chemotherapy (T3) | Patient 3-6 Months After the Completion of Therapy (T5) | Parent 3-6 Months After the Completion of Therapy (T5)
Number analyzed (Participants) | 142 | 142 | 128 | 128 | 103 | 103
units on a scale | 71.3 (27.9) | 70.3 (27.9) | 73.8 (27.7) | 63.2 (29.6) | 78.5 (25.4) | 72.7 (28.1)
Statistical Analysis 1: Comparison: Patient Completion of 2 Cycles of Chemotherapy (T2) vs Parent Completion of 2 Cycles of Chemotherapy (T2); Test type: Superiority or Other; p = 0.4263, Wilcoxon signed rank test
Statistical Analysis 2: Comparison: Patient Completion of 2 Cycles of Chemotherapy (T2) vs Parent Completion of 2 Cycles of Chemotherapy (T2); Test type: Superiority or Other; p < 0.0001, Spearman Correlation Coefficients; Spearman Correlation Coefficients = 0.51
Statistical Analysis 3: Comparison: Patient Completion of 4 Cycles of Chemotherapy (T3) vs Parent Completion of 4 Cycles of Chemotherapy (T3); Test type: Superiority or Other; p < 0.0001, Wilcoxon signed rank test
Statistical Analysis 4: Comparison: Patient Completion of 4 Cycles of Chemotherapy (T3) vs Parent Completion of 4 Cycles of Chemotherapy (T3); Test type: Superiority or Other; p < 0.0001, Spearman Correlation Coefficients; Spearman Correlation Coefficients = 0.54
Statistical Analysis 5: Comparison: Patient 3-6 Months After the Completion of Therapy (T5) vs Parent 3-6 Months After the Completion of Therapy (T5); Test type: Superiority or Other; p = 0.0468, Wilcoxon signed rank test
Statistical Analysis 6: Comparison: Patient 3-6 Months After the Completion of Therapy (T5) vs Parent 3-6 Months After the Completion of Therapy (T5); Test type: Superiority or Other; p < 0.0001, Spearman Correlation Coefficients; Spearman Correlation Coefficients = 0.55

11. Secondary Outcome: Correlation of Agreement Between Patient Treatment Anxiety QoL and Parent Proxy Treatment Anxiety QoL at Multiple Time Points.
Description: Assess and compare the patient reported and parent proxy treatment anxiety quality of life across multiple time points using the Peds Quality of Life version 3. Assessment was performed across all risk groups. The QL scoring is a 5-point Likert scale from 0 (never) to 4 (almost always). Scores are transformed on a scale from 0 to 100. Items are reverse scored and linearly transformed to a 0-100 scale as follows: 0=100, 1=75, 2=50, 3=25, and 4=0. Total score is the sum of all items over the number of items answered on all scales. The higher the score, the better the quality of life.
Time Frame: as for outcome 8
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patient Completion of 2 Cycles of Chemotherapy (T2) | Parent Completion of 2 Cycles of Chemotherapy (T2) | Patient Completion of 4 Cycles of Chemotherapy (T3) | Parent Completion of 4 Cycles of Chemotherapy (T3) | Patient 3-6 Months After the Completion of Therapy (T5) | Parent 3-6 Months After the Completion of Therapy (T5)
Number analyzed (Participants) | 140 | 140 | 130 | 130 | 104 | 104
units on a scale | 84.1 (20.6) | 72.8 (25.2) | 82.8 (22.7) | 71.1 (24.9) | 82.1 (23) | 77.6 (24.2)
Statistical Analysis 1: Comparison: Patient Completion of 2 Cycles of Chemotherapy (T2) vs Parent Completion of 2 Cycles of Chemotherapy (T2); Test type: Superiority or Other; p < 0.0001, Wilcoxon signed rank test
Statistical Analysis 2: Comparison: Patient Completion of 2 Cycles of Chemotherapy (T2) vs Parent Completion of 2 Cycles of Chemotherapy (T2); Test type: Superiority or Other; p = 0.0019, Spearman Correlation Coefficients; Spearman Correlation Coefficients = 0.26
Statistical Analysis 3: Comparison: Patient Completion of 4 Cycles of Chemotherapy (T3) vs Parent Completion of 4 Cycles of Chemotherapy (T3); Test type: Superiority or Other; p < 0.0001, Wilcoxon signed rank test
Statistical Analysis 4: Comparison: Patient Completion of 4 Cycles of Chemotherapy (T3) vs Parent Completion of 4 Cycles of Chemotherapy (T3); Test type: Superiority or Other; p = 0.0704, Spearman Correlation Coefficients; Spearman Correlation Coefficients = 0.16
Statistical Analysis 5: Comparison: Patient 3-6 Months After the Completion of Therapy (T5) vs Parent 3-6 Months After the Completion of Therapy (T5); Test type: Superiority or Other; p = 0.0200, Wilcoxon signed rank test
Statistical Analysis 6: Comparison: Patient 3-6 Months After the Completion of Therapy (T5) vs Parent 3-6 Months After the Completion of Therapy (T5); Test type: Superiority or Other; p < 0.0001, Spearman Correlation Coefficients; Spearman Correlation Coefficients = 0.42

12. Secondary Outcome: Correlation of Agreement Between Patient Worry QoL and Parent Proxy Worry QoL at Multiple Time Points.
Description: Assess and compare the patient reported and parent proxy worry quality of life across multiple time points using the Peds Quality of Life version 3. Assessment was performed across all risk groups. The QL scoring is a 5-point Likert scale from 0 (never) to 4 (almost always). Scores are transformed on a scale from 0 to 100. Items are reverse scored and linearly transformed to a 0-100 scale as follows: 0=100, 1=75, 2=50, 3=25, and 4=0. Total score is the sum of all items over the number of items answered on all scales. The higher the score, the better the quality of life.
Time Frame: as for outcome 8
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patient Completion of 2 Cycles of Chemotherapy (T2) | Parent Completion of 2 Cycles of Chemotherapy (T2) | Patient Completion of 4 Cycles of Chemotherapy (T3) | Parent Completion of 4 Cycles of Chemotherapy (T3) | Patient 3-6 Months After the Completion of Therapy (T5) | Parent 3-6 Months After the Completion of Therapy (T5)
Number analyzed (Participants) | 141 | 141 | 131 | 131 | 101 | 101
units on a scale | 64.5 (24.2) | 64.5 (21.3) | 64.7 (24.9) | 64.7 (23.6) | 67.1 (28) | 68.6 (25.9)
Statistical Analysis 1: Comparison: Patient Completion of 2 Cycles of Chemotherapy (T2) vs Parent Completion of 2 Cycles of Chemotherapy (T2); Test type: Superiority or Other; p = 0.7192, Wilcoxon signed rank test
Statistical Analysis 2: Comparison: Patient Completion of 2 Cycles of Chemotherapy (T2) vs Parent Completion of 2 Cycles of Chemotherapy (T2); Test type: Superiority or Other; p < 0.0001, Spearman Correlation Coefficients; Spearman Correlation Coefficients = 0.42
Statistical Analysis 3: Comparison: Patient Completion of 4 Cycles of Chemotherapy (T3) vs Parent Completion of 4 Cycles of Chemotherapy (T3); Test type: Superiority or Other; p = 0.8663, Wilcoxon signed rank test
Statistical Analysis 4: Comparison: Patient Completion of 4 Cycles of Chemotherapy (T3) vs Parent Completion of 4 Cycles of Chemotherapy (T3); Test type: Superiority or Other; p < 0.0001, Spearman Correlation Coefficients; Spearman Correlation Coefficients = 0.41
Statistical Analysis 5: Comparison: Patient 3-6 Months After the Completion of Therapy (T5) vs Parent 3-6 Months After the Completion of Therapy (T5); Test type: Superiority or Other; p = 0.7626, Wilcoxon signed rank test
Statistical Analysis 6: Comparison: Patient 3-6 Months After the Completion of Therapy (T5) vs Parent 3-6 Months After the Completion of Therapy (T5); Test type: Superiority or Other; p < 0.0001, Spearman Correlation Coefficients; Spearman Correlation Coefficients = 0.58

13. Secondary Outcome: Correlation of Agreement Between Patient Cognitive Problems (Child + Teen) QoL and Parent Proxy Cognitive Problems (Child + Teen) QoL at Multiple Time Points.
Description: Assess and compare the patient reported and parent proxy cognitive problems (child + teen) quality of life across multiple time points using the Peds Quality of Life version 3. Assessment was performed across all risk groups. The QL scoring is a 5-point Likert scale from 0 (never) to 4 (almost always). Scores are transformed on a scale from 0 to 100. Items are reverse scored and linearly transformed to a 0-100 scale as follows: 0=100, 1=75, 2=50, 3=25, and 4=0. Total score is the sum of all items over the number of items answered on all scales. The higher the score, the better the quality of life.
Time Frame: as for outcome 8
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patient Completion of 2 Cycles of Chemotherapy (T2) | Parent Completion of 2 Cycles of Chemotherapy (T2) | Patient Completion of 4 Cycles of Chemotherapy (T3) | Parent Completion of 4 Cycles of Chemotherapy (T3) | Patient 3-6 Months After the Completion of Therapy (T5) | Parent 3-6 Months After the Completion of Therapy (T5)
Number analyzed (Participants) | 139 | 139 | 126 | 126 | 105 | 105
units on a scale | 77.6 (19.2) | 75.7 (19.7) | 78.9 (20.2) | 74.3 (22.2) | 80.8 (20.4) | 76.3 (22.6)
Statistical Analysis 1: Comparison: Patient Completion of 2 Cycles of Chemotherapy (T2) vs Parent Completion of 2 Cycles of Chemotherapy (T2); Test type: Superiority or Other; p = 0.4807, Wilcoxon signed rank test
Statistical Analysis 2: Comparison: Patient Completion of 2 Cycles of Chemotherapy (T2) vs Parent Completion of 2 Cycles of Chemotherapy (T2); Test type: Superiority or Other; p < 0.0001, Spearman Correlation Coefficients; Spearman Correlation Coefficients = 0.36
Statistical Analysis 3: Comparison: Patient Completion of 4 Cycles of Chemotherapy (T3) vs Parent Completion of 4 Cycles of Chemotherapy (T3); Test type: Superiority or Other; p = 0.0824, Wilcoxon signed rank test
Statistical Analysis 4: Comparison: Patient Completion of 4 Cycles of Chemotherapy (T3) vs Parent Completion of 4 Cycles of Chemotherapy (T3); Test type: Superiority or Other; p < 0.0001, Spearman Correlation Coefficients; Spearman Correlation Coefficients = 0.39
Statistical Analysis 5: Comparison: Patient 3-6 Months After the Completion of Therapy (T5) vs Parent 3-6 Months After the Completion of Therapy (T5); Test type: Superiority or Other; p = 0.0496, Wilcoxon signed rank test
Statistical Analysis 6: Comparison: Patient 3-6 Months After the Completion of Therapy (T5) vs Parent 3-6 Months After the Completion of Therapy (T5); Test type: Superiority or Other; p < 0.0001, Spearman Correlation Coefficients; Spearman Correlation Coefficients = 0.50

14. Secondary Outcome: Correlation of Agreement Between Patient Perceived Physical Appearance QoL and Parent Proxy Perceived Physical Appearance QoL at Multiple Time Points.
Description: Assess and compare the patient reported and parent proxy perceived physical appearance quality of life across multiple time points using the Peds Quality of Life version 3. Assessment was performed across all risk groups. The QL scoring is a 5-point Likert scale from 0 (never) to 4 (almost always). Scores are transformed on a scale from 0 to 100. Items are reverse scored and linearly transformed to a 0-100 scale as follows: 0=100, 1=75, 2=50, 3=25, and 4=0. Total score is the sum of all items over the number of items answered on all scales. The higher the score, the better the quality of life.
Time Frame: as for outcome 8
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patient Completion of 2 Cycles of Chemotherapy (T2) | Parent Completion of 2 Cycles of Chemotherapy (T2) | Patient Completion of 4 Cycles of Chemotherapy (T3) | Parent Completion of 4 Cycles of Chemotherapy (T3) | Patient 3-6 Months After the Completion of Therapy (T5) | Parent 3-6 Months After the Completion of Therapy (T5)
Number analyzed (Participants) | 143 | 143 | 126 | 126 | 105 | 105
units on a scale | 77.5 (23.1) | 71.9 (25.9) | 77.6 (23.3) | 71.2 (26.6) | 78.4 (25) | 80.5 (22.8)
Statistical Analysis 1: Comparison: Patient Completion of 2 Cycles of Chemotherapy (T2) vs Parent Completion of 2 Cycles of Chemotherapy (T2); Test type: Superiority or Other; p = 0.0157, Wilcoxon signed rank test
Statistical Analysis 2: Comparison: Patient Completion of 2 Cycles of Chemotherapy (T2) vs Parent Completion of 2 Cycles of Chemotherapy (T2); Test type: Superiority or Other; p < 0.0001, Spearman Correlation Coefficients; Spearman Correlation Coefficients = 0.37
Statistical Analysis 3: Comparison: Patient Completion of 4 Cycles of Chemotherapy (T3) vs Parent Completion of 4 Cycles of Chemotherapy (T3); Test type: Superiority or Other; p = 0.0014, Wilcoxon signed rank test
Statistical Analysis 4: Comparison: Patient Completion of 4 Cycles of Chemotherapy (T3) vs Parent Completion of 4 Cycles of Chemotherapy (T3); Test type: Superiority or Other; p < 0.0001, Spearman Correlation Coefficients; Spearman Correlation Coefficients = 0.43
Statistical Analysis 5: Comparison: Patient 3-6 Months After the Completion of Therapy (T5) vs Parent 3-6 Months After the Completion of Therapy (T5); Test type: Superiority or Other; p = 0.1478, Wilcoxon signed rank test
Statistical Analysis 6: Comparison: Patient 3-6 Months After the Completion of Therapy (T5) vs Parent 3-6 Months After the Completion of Therapy (T5); Test type: Superiority or Other; p < 0.0001, Spearman Correlation Coefficients; Spearman Correlation Coefficients = 0.56

15. Secondary Outcome: Correlation of Agreement Between Patient Communication QoL and Parent Proxy Communication QoL at Multiple Time Points.
Description: Assess and compare the patient reported and parent proxy communication quality of life across multiple time points using the Peds Quality of Life version 3. Assessment was performed across all risk groups. The QL scoring is a 5-point Likert scale from 0 (never) to 4 (almost always). Scores are transformed on a scale from 0 to 100. Items are reverse scored and linearly transformed to a 0-100 scale as follows: 0=100, 1=75, 2=50, 3=25, and 4=0. Total score is the sum of all items over the number of items answered on all scales. The higher the score, the better the quality of life.
Time Frame: as for outcome 8
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patient Completion of 2 Cycles of Chemotherapy (T2) | Parent Completion of 2 Cycles of Chemotherapy (T2) | Patient Completion of 4 Cycles of Chemotherapy (T3) | Parent Completion of 4 Cycles of Chemotherapy (T3) | Patient 3-6 Months After the Completion of Therapy (T5) | Parent 3-6 Months After the Completion of Therapy (T5)
Number analyzed (Participants) | 142 | 142 | 127 | 127 | 105 | 105
units on a scale | 78.3 (19.5) | 73.6 (27.8) | 80.6 (19.9) | 74.9 (25.2) | 83.7 (19.5) | 83.1 (20.6)
Statistical Analysis 1: Comparison: Patient Completion of 2 Cycles of Chemotherapy (T2) vs Parent Completion of 2 Cycles of Chemotherapy (T2); Test type: Superiority or Other; p = 0.0831, Wilcoxon signed rank test
Statistical Analysis 2: Comparison: Patient Completion of 2 Cycles of Chemotherapy (T2) vs Parent Completion of 2 Cycles of Chemotherapy (T2); Test type: Superiority or Other; p = 0.0027, Spearman Correlation Coefficients; Spearman Correlation Coefficients = 0.25
Statistical Analysis 3: Comparison: Patient Completion of 4 Cycles of Chemotherapy (T3) vs Parent Completion of 4 Cycles of Chemotherapy (T3); Test type: Superiority or Other; p = 0.0135, Wilcoxon signed rank test
Statistical Analysis 4: Comparison: Patient Completion of 4 Cycles of Chemotherapy (T3) vs Parent Completion of 4 Cycles of Chemotherapy (T3); Test type: Superiority or Other; p = 0.0024, Spearman Correlation Coefficients; Spearman Correlation Coefficients = 0.27
Statistical Analysis 5: Comparison: Patient 3-6 Months After the Completion of Therapy (T5) vs Parent 3-6 Months After the Completion of Therapy (T5); Test type: Superiority or Other; p = 0.9848, Wilcoxon signed rank test
Statistical Analysis 6: Comparison: Patient 3-6 Months After the Completion of Therapy (T5) vs Parent 3-6 Months After the Completion of Therapy (T5); Test type: Superiority or Other; p = 0.0974, Spearman Correlation Coefficients; Spearman Correlation Coefficients = 0.16

16. Secondary Outcome: Correlation of Agreement Between Patient PedsQL3 (Composite) QoL and Parent Proxy PedsQL3 (Composite) QoL at Multiple Time Points.
Description: Assess and compare the patient reported and parent proxy PedsQL3 (composite) quality of life across multiple time points using the Peds Quality of Life version 3. Assessment was performed across all risk groups. The QL scoring is a 5-point Likert scale from 0 (never) to 4 (almost always). Scores are transformed on a scale from 0 to 100. Items are reverse scored and linearly transformed to a 0-100 scale as follows: 0=100, 1=75, 2=50, 3=25, and 4=0. Total score is the sum of all items over the number of items answered on all scales. The higher the score, the better the quality of life.
Time Frame: as for outcome 8
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patient Completion of 2 Cycles of Chemotherapy (T2) | Parent Completion of 2 Cycles of Chemotherapy (T2) | Patient Completion of 4 Cycles of Chemotherapy (T3) | Parent Completion of 4 Cycles of Chemotherapy (T3) | Patient 3-6 Months After the Completion of Therapy (T5) | Parent 3-6 Months After the Completion of Therapy (T5)
Number analyzed (Participants) | 132 | 132 | 118 | 118 | 91 | 91
units on a scale | 72.4 (14.6) | 68.3 (14.7) | 72.7 (16.7) | 67.6 (16.3) | 78.1 (16) | 77.6 (16)
Statistical Analysis 1: Comparison: Patient Completion of 2 Cycles of Chemotherapy (T2) vs Parent Completion of 2 Cycles of Chemotherapy (T2); Test type: Superiority or Other; p = 0.0040, Wilcoxon signed rank test
Statistical Analysis 2: Comparison: Patient Completion of 2 Cycles of Chemotherapy (T2) vs Parent Completion of 2 Cycles of Chemotherapy (T2); Test type: Superiority or Other; p < 0.0001, Spearman Correlation Coefficients; Spearman Correlation Coefficients = 0.43
Statistical Analysis 3: Comparison: Patient Completion of 4 Cycles of Chemotherapy (T3) vs Parent Completion of 4 Cycles of Chemotherapy (T3); Test type: Superiority or Other; p = 0.0012, Wilcoxon signed rank test
Statistical Analysis 4: Comparison: Patient Completion of 4 Cycles of Chemotherapy (T3) vs Parent Completion of 4 Cycles of Chemotherapy (T3); Test type: Superiority or Other; p < 0.0001, Spearman Correlation Coefficients; Spearman Correlation Coefficients = 0.54
Statistical Analysis 5: Comparison: Patient 3-6 Months After the Completion of Therapy (T5) vs Parent 3-6 Months After the Completion of Therapy (T5); Test type: Superiority or Other; p = 0.8108, Wilcoxon signed rank test
Statistical Analysis 6: Comparison: Patient 3-6 Months After the Completion of Therapy (T5) vs Parent 3-6 Months After the Completion of Therapy (T5); Test type: Superiority or Other; p < 0.0001, Spearman Correlation Coefficients; Spearman Correlation Coefficients = 0.55

17. Other Pre Specified Outcome: Event-free Survival Probability by Risk Group at 10-year Follow-Up
Description: Event-free survival (EFS) is based on the time from protocol enrollment to the occurrence of first event (relapse or progressive disease, subsequent malignancy, or death from any cause). Patients not experiencing an event are censored at their last follow-up date. Event-free Survival Probability will be estimated by Kaplan-Meier (KM) method with a 95% confidence interval calculated using the with Greenwood's formula.
Time Frame: 10-year follow-up after protocol enrollment
Population: Nine patients were ineligible for analysis.
Measure: Number (95% Confidence Interval); unit: probability 10 yr. event free survival
Arm/Group | Favorable Risk | Intermediate Risk | Unfavorable Risk, Group 1 | Unfavorable Risk, Group 2
Number analyzed (Participants) | 88 | 46 | 12 | 141
probability 10 yr. event free survival | 0.874 [0.805 to 0.944] | 0.844 [0.739 to 0.950] | 0.667 [0.400 to 0.933] | 0.785 [0.716 to 0.853]
Statistical Analysis 1: Comparison: Favorable Risk; Test type: Superiority or Other; KM Event-free survival estimate = 0.874, 95% CI 2-sided [0.805 to 0.944]
Statistical Analysis 2: Comparison: Intermediate Risk; Test type: Superiority or Other; KM event-free survival estimate = 0.844, 95% CI 2-sided [0.739 to 0.950]
Statistical Analysis 3: Comparison: Unfavorable Risk, Group 1; Test type: Superiority or Other; KM event-free survival estimate = 0.667, 95% CI 2-sided [0.400 to 0.933]
Statistical Analysis 4: Comparison: Unfavorable Risk, Group 2; Test type: Superiority or Other; KM event-free survival estimate = 0.785, 95% CI 2-sided [0.716 to 0.853]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the date a patient went on study through the completion of therapy. The elapsed timeframe for adverse event collection was eleven years (March, 2000 through May, 2011).
Arm/Group | Favorable Risk | Intermediate Risk | Unfavorable Risk, Group 1 | Unfavorable Risk, Group 2
Serious Adverse Events (participants affected / at risk) | 0/91 | 0/46 | 0/13 | 1/146
Other Adverse Events (participants affected / at risk) | 54/88 | 39/46 | 12/13 | 116/146
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Favorable Risk (N=91) | Intermediate Risk (N=46) | Unfavorable Risk, Group 1 (N=13) | Unfavorable Risk, Group 2 (N=146)
Thrombosis/thrombus/embolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Favorable Risk (N=88) | Intermediate Risk (N=46) | Unfavorable Risk, Group 1 (N=13) | Unfavorable Risk, Group 2 (N=146)
Hemoglobin (Blood and lymphatic system disorders) | 0 (0) | 2 (3) | 1 (4) | 52 (85)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 15 (22) | 24 (51) | 10 (42) | 89 (236)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 24 (66)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 53 (118) | 39 (98) | 11 (51) | 101 (234)
Platelets (Blood and lymphatic system disorders) | 0 (0) | 3 (5) | 1 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mucositis/stomatitis (functional/symptomatic), Oral cavity (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 4 (4) | 1 (1) | 0 (0)
Febrile neutropenia (fever of unknown origin without clinically or microbiologically documented infe (Infections and infestations) | 0 (0) | 7 (7) | 2 (2) | 12 (13)
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC<1.0x10e (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infection with unknown ANC, Blood (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 7 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes